CLINICAL TRIAL: NCT05116007
Title: Phase Ib Clinical Study of Anti-PD-1 and VEGF Bispecific Antibody AK112 in Combination With Etoposide and Carboplatin for the First-line Treatment of Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: Anti-PD-1 and VEGF Bispecific Antibody AK112 in Combination With Chemotherapy in Patients With ES-SCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK112-103
Record Dates: First submitted 2021-09-21; First posted 2021-11-10 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: SCLC, Extensive Stage
MeSH Terms: interventions — Etoposide; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Subjects receive AK112 plus Etoposide and Carboplatin every 3- week cycle (Q3W) for 4 cycles followed by AK112 until progression.
  Interventions: Drug: AK112; Drug: Etoposide; Drug: Carboplatin

INTERVENTIONS:
Drug: AK112 — IV infusion
Drug: Etoposide — Etoposide intravenous infusion was administered at a dose of 100 mg/m^2 on Days 1, 2, and 3 of each 21-day cycle during the induction phase (Cycles 1-4).
Drug: Carboplatin — Carboplatin intravenous infusion to achieve an initial target AUC of 5 mg/mL/min was administered on Day 1 of each 21-day cycle during the induction phase (Cycles 1-4)

SUMMARY:
Phase Ib open label, multicenter study to evaluate the efficacy and safety of anti-PD-1 and VEGF bispecific antibody (AK112) combined with chemotherapy in patients with ES-SCLC.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) is an aggressive type of neuroendocrine tumor with the majority of patients (about 60-70%) being diagnosed with metastatic disease and with a median survival ranging from 7 to 12 months. Combination chemotherapy , namely a platinum and etoposide-based regimen, represents the cornerstone of treatment for extensive stage SCLC(ES-SCLC). Despite this the duration of response is short and nearly all patients develop disease relapse or progression. The recent approval of atezolizumab in combination with carboplatin and etoposide as first line in patients with ES- SCLC is surely a step forward in the understanding the molecular landscape and treatment of this complex tumor, but new therapeutic approaches need to be explored.This trial aims to assess the safety and efficacy of a new therapeutic strategy that combines to carboplatin and etoposide, and a new drug AK112.The treatment will start with an induction phase during which eligible patients will receive, by intravenous way, a combination of the above mentioned drugs according to a specific administration regimen. This phase will last about 12 weeks. Thereafter the treatment will proceed with a maintenence phase lasting for a maximum of 24 months during which the patients will receive only AK112, by intravenous way. Treatment will be discontnued in case of until the toxicity became intolerable, the investigator determined that there was no further clinical benefit (based on a combination of RECIST V1.1 imaging assessment and clinical status), 24 months of treatment was completed, or the study was withdrawn for other reasons. During the study period the patients will undergo to periodic visits and laboratory, radiologic assessments to monitor the efficacy and the safety of the ongoing treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old (at the time of inform consent obtained).
* Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures).
* Histologically or cytologically confirmed ES-SCLC (per the Veterans Administration Lung Study Group [VALG] staging system).
* Be able to provide formalin fixed, paraffin-embedded (FFPE) tumor tissue obtained from either a core or excisional tumor biopsy.
* Have a life expectancy of at least 3 months.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by investigator
* Has adequate organ function
* All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.

Exclusion Criteria:

* Undergone major surgery within 30 days prior to the first dose of study treatment
* History of prior malignancy except that basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Active central nervous system (CNS) metastases
* History of active autoimmune disease that has required systemic treatment in the past 2 years (i.e.,corticosteroids or immunosuppressive drugs).
* Active infection requiring systemic therapy
* Active Hepatitis B or Hepatitis C
* History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 12 months prior to day 1 of study treatment;
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Grade 3 or higher adverse events (AEs) | Interval between the date of enrollment and the date of death from any cause, up to a maximum of 2 years
  Frequency and severity of adverse events measured according to NCI Common Toxicity Criteria Adverse Event (CTCAE), version 5.0
Objective Response Rate (ORR) | Interval between the date of enrollment and the date of death from any cause, up to a maximum of 18 months.
  ORR is proportion of subjects with complete response(CR) or partial response(PR). Tumor responses will be evaluated according to RECIST 1.1 criteria. Patients with no tumor assessment after baseline will be classified as non-responders.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Interval between the date of enrollment and the date of death due to any cause , up to a maximum of approximately 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST V1.1
Progression free survival (PFS) | Interval between the date of enrollment and the date of progressive disease, or death due to any cause (whichever occurs first), up to a maximum of 24 months.
  PFS is defined as the time from the date of first dosing till the first documentation of disease progression (per RECIST v1.1) assessed by the investigator or death due to any cause (whichever occurs first)
Overall survival (OS) | Interval between the date of enrollment and the date of death from any cause, up to a maximum of 24 months.
  OS is the time from the date of randomization or first dosing date to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, Professor, Principal Investigator — Shanghai Lung Cancer Center, Shanghai Chest Hospital, Shanghai Jiaotong University, P. R. China
Locations (1):
- Shun Lu, Shanghai, Shanghai Municipality, China